CLINICAL TRIAL: NCT00341484
Title: Genetic Susceptibility to Oncogenic Viruses
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999998026; OH98-C-N026
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Liver Neoplasms; HIV Infections
Keywords: Genetics; Liver Cancer; HIV
MeSH Terms: conditions — Liver Neoplasms; HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
An NCI goal is to identify every human gene that predisposes people to cancer. Recent studies of HIV-1 indicate that genetic polymorphisms can affect susceptibility to viral infections and that such alleles may be racially restricted, a range of racial and ethnic groups should be included in such studies. We propose to examine genetic determinants of infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) in an ethnically diverse population of injection drug users (IDUs). HBV and HCV are important causes of hepatocellular carcinoma, but little is known about genetic factors that alter susceptibility to these infections. Subjects will be recruited in diverse inner-city neighborhoods as part of the University of California, San Francisco's Urban Health Study. Since 1986, this study has successfully recruited and evaluated IDUs from street-based settings. About half of the participants are African-American, one-third are white, 10% are Latino, and the remainder are Asian or Native American. The mean duration of drug use exceeds 20 years. About 80% of subjects have evidence of HBV infection and a similar prevalence of HCV infections is anticipated. We will enroll about 1500 subjects over a 13 month period. Archived, unlinked serum specimens may be obtained from previous enrollees to increase the sample size, as needed. Highly exposed-uninfected subjects will be ascertained on the basis of the serologic testing for each virus, as well as the duration and frequency of injection drug use. These highly exposed-uninfected subjects will be compared to infected subjects with regard to their frequency of genetic polymorphisms (chemokines, chemokine receptors, human leukocyte antigens, and others), in collaboration with scientists from NCI's Laboratory of Genomic Diversity.

DETAILED DESCRIPTION:
An NCI goal is to identify every human gene that predisposes people to cancer. Recent studies of HIV -1 indicate that genetic polymorphisms can affect susceptibility to viral infections and that such alleles may be detected in studies of small numbers of highly exposed-uninfected subjects. Because such alleles may be racially restricted, a range of racial and ethnic groups should be included in such studies. We propose to examine genetic determinants of infection with hepatitis B virus (HBV) and hepatitis C virus (HCV) in an ethnically diverse population of injection drug users (lDUs). HBV and HCV are important causes of hepatocellular carcinoma, but little is known about genetic factors that alter susceptibility to these infections. Subjects will be recruited in diverse inner-city neighborhoods as part of the University of California, San Francisco's Urban Health Study. Since 1986, this study has successfully recruited and evaluated IDUs from street-based settings. About half of the participants are African-American, one-third are white, 10% are Latino, and the remainder are Asian or Native American. The mean duration of drug use exceeds 20 years. About 80% of subjects have evidence of HBV infection and a similar prevalence of HCV infection is anticipated. We will enroll about 1500 subjects over a 13 month period. Archived, unlinked serum specimens may obtained from previous enrollees to increase the sample size, as needed. Highly exposed-uninfected subjects will be ascertained on the basis of the serologic testing for each virus, as well as the duration and frequency of injection drug use. These highly exposed-uninfected subjects will be compared to infected subjects with regard to their frequency of genetic polymorphisms (chemokines, chemokine receptors, human leukocyte antigens, and others), in collaboration with scientists from NCI's Laboratory of Genomic Diversity.

ELIGIBILITY:
* INCLUSION CRITERIA:

  18 years or older

Active IDU as verified by self-report and physical examination for visible signs consistent with multiple drug injection.

EXCLUSION CRITERIA:

Subject unable to give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of inner-city neighborhoods in San Francisco, CA.
Sampling Method: Non-Probability Sample
Enrollment: 2580 (Actual)
Dates: Start 1998-06-01 (Actual); Primary Completion 2007-06-05 (Actual); Study Completion 2007-06-05 (Actual)

PRIMARY OUTCOMES:
Genetic determinants | 5 years
  genetic determinants

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R O'Brien, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Aka PV, Kuniholm MH, Pfeiffer RM, Wang AS, Tang W, Chen S, Astemborski J, Plankey M, Villacres MC, Peters MG, Desai S, Seaberg EC, Edlin BR, Strickler HD, Thomas DL, Prokunina-Olsson L, Sharp GB, O'Brien TR. Association of the IFNL4-DeltaG Allele With Impaired Spontaneous Clearance of Hepatitis C Virus. J Infect Dis. 2014 Feb 1;209(3):350-4. doi: 10.1093/infdis/jit433. Epub 2013 Aug 15. PMID 23956438
- [Background] Prokunina-Olsson L, Muchmore B, Tang W, Pfeiffer RM, Park H, Dickensheets H, Hergott D, Porter-Gill P, Mumy A, Kohaar I, Chen S, Brand N, Tarway M, Liu L, Sheikh F, Astemborski J, Bonkovsky HL, Edlin BR, Howell CD, Morgan TR, Thomas DL, Rehermann B, Donnelly RP, O'Brien TR. A variant upstream of IFNL3 (IL28B) creating a new interferon gene IFNL4 is associated with impaired clearance of hepatitis C virus. Nat Genet. 2013 Feb;45(2):164-71. doi: 10.1038/ng.2521. Epub 2013 Jan 6. PMID 23291588
- [Background] Uccellini L, Tseng FC, Monaco A, Shebl FM, Pfeiffer R, Dotrang M, Buckett D, Busch MP, Wang E, Edlin BR, Marincola FM, O'Brien TR. HCV RNA levels in a multiethnic cohort of injection drug users: human genetic, viral and demographic associations. Hepatology. 2012 Jul;56(1):86-94. doi: 10.1002/hep.25652. Epub 2012 Jun 1. PMID 22331649